CLINICAL TRIAL: NCT05596747
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3209590 Following Multiple Weekly Doses in Chinese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3209590 in Chinese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18221; I8H-MC-BDDC (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY3209590 (Experimental): LY3209590 administered subcutaneously (SC).
  Interventions: Drug: LY3209590
- Insulin glargine (Active Comparator): Insulin glargine administered SC.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: LY3209590 — Administered SC.
  Arms: LY3209590
Drug: Insulin Glargine — Administered SC.
  Arms: Insulin glargine

SUMMARY:
The main purpose of this study is to evaluate the safety of a study drug known as LY3209590 in Chinese participants with type 2 diabetes mellitus who are on a stable dose of basal insulin. Side effects and tolerability will be documented. Blood samples will be taken to assess how the body processes the study drug and the effect of the study drug on blood sugar levels. The study will last up to 18 weeks and may include 18 visits for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Type 2 Diabetes Mellitus (T2DM) and treated with basal insulin and up to one non-insulin anti-hyperglycemic medication.
* Body mass index (BMI) of 18.5 to 40.0 kilograms per meter squared (kg/m²)
* Have received a stable daily dose of basal insulin at screening
* Have hemoglobin A1c (HbA1c) greater than or equal to (≥)6.5 percent (%) and less than or equal to (≤)10.0% at screening
* Native Chinese participant who has both parents and all 4 grandparents of Chinese origin.

Exclusion Criteria:

* Have a diagnosis of type 1 diabetes mellitus or latent autoimmune diabetes
* Have a history of ketoacidosis or hyperosmolar state/coma episode or severe hypoglycemia or hypoglycemia unawareness in the 6 months prior to screening
* Are receiving insulin other than once daily basal insulin
* Have any active infectious or serious disease or major organs insufficiency
* Women who are pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events (AEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 12
  Number of Participants with One or More AEs and SAEs Considered by the Investigator to be Related to Study Drug Administration
Incidence and Severity of Hypoglycemia | Baseline up to Week 12
  Incidence and Severity of Hypoglycemia

SECONDARY OUTCOMES:
Pharmacodynamics (PD): Change from Baseline in Fasting Plasma Glucose | Baseline through Week 6
  PD: Change from Baseline in Fasting Plasma Glucose
PD: Change from Baseline in 7-Point Glucose | Baseline through Week 6
  PD: Change from Baseline in 7-Point Glucose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No